CLINICAL TRIAL: NCT05801289
Title: Quetiapine as a Prophylactic Agent for Early Postoperative Delirium in High Risk Patients in Open Heart Surgeries
Brief Title: Quetiapine as Prophylaxis for Delirium in CABG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R 293/2022
Record Dates: First submitted 2023-02-22; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Q (Active Comparator): will receive 25 mg quetiapine at night of surgery and 25 mg daily for 7 days postoperative
  Interventions: Drug: Quetiapine
- Group C (No Intervention): will receive placebo alone

INTERVENTIONS:
Drug: Quetiapine — Giving the drug to group Q
  Other Names: Seroquel
  Arms: Group Q

SUMMARY:
low-dose quetiapine may be effective in preventing delirium in patients. The purpose of this study is to evaluate the efficacy and safety of quetiapine for delirium prophylaxis in cabg

DETAILED DESCRIPTION:
Group Q: will receive 25 mg quetiapine at night of surgery and 25 mg daily for 7 days postoperative (30 patients).

Group C: will receive placebo alone (30 patients). During the study period, enrolled patients will be assessed for delirium once daily (from 7:00 AM to 7:00 PM), and the assessment will be performed in two steps. First, level of sedation will be assessed using the RASS. If the patient will be deeply sedated or unarousable (RASS -4 or -5), the assessment will not be performed and the patient will be reassessed at a later time. If the patient has a RASS of -3to +4, then the assessment will be continued to the next step.

Second, delirium will be diagnosed using the CAM-ICU. The screening tool detects four features of delirium: acute onset of mental status change or a ﬂuctuating course, inattention, disorganized thinking, and altered level of consciousness. To have delirium diagnosed, a patient displays the ﬁrst two features with either the third or fourth feature.

The primary outcome is delirium incidence diagnosed with the CAM_ICU within the study period. If the CAM_ICU is positive at least once during the study period, it will be recorded that a delirium occurred.

Secondary outcomes is the rate of positive CAM-ICU (the number of positive CAM-ICU counts/the number of total CAM-ICU counts), days without delirium (number of days from the start of treatment until delirium), the duration of delirium if it appear (number of days with delirium), severity of delirium as measured with delirium rating scale revised 98 (DRS-R-89), the length of stay in the ICU, the length of stay in the hospital, the duration of intubation, a successful extubation, the ICU mortality, the overall mortality, measurement of QTc prolongation, and the use of rescue medication.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 65 or older old of age undergoing open heart surgery and having an equal or greater score of 5 on the scale of Delphi.

* Age: 70-79 years: 1 point; ≥ 80 years: 2 points
* Physical activity: need for assistance, not self-sufficient: 2 points
* Alcoholism: 1 point
* Hearing impaired: 1 point
* History of delirium: 2 points
* Emergency of surgery: 2 points
* No laparoscopic surgery: 2 points
* Admission critical unites: 3 points
* Value of C reactive protein (CRP) ≥ 10mg/dl: 1 point

Exclusion Criteria:

.Patient refusal.

* Allergy to quetiapine
* Patients with a score less than 5 on Delphi scale
* Diagnosis of delirium on admission initial CAM-ICU (the Confusion Assessment Method-ICU) positive)
* Could not communicate due to previously diagnosed irreversible neurologic disease (stroke, cerebral hemorrhage, traumatic brain injury, dementia, etc.)
* High risk for ventricular arrhythmias (Corrected QT interval ≥ 460 millisecond in men, ≥ 470 millisecond in women or ongoing treatment with drugs known to prolong the QT interval (e.g., erythromycin, class Ia, Ic, III anti-arrhythmic drugs)
* Second or third degree heart block
* High risk for drug interaction with quetiapine (phenytoin, carbamazepine, barbiturates)
* Electrolyte disturbance : Potassium less than 3 or magnesium less than 1.5
* Patient on antipsychotic drug treatment prior to admission
* Parkinson's disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-04 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
delirium incidence | 3 days postoperative
  CAM_ICU

SECONDARY OUTCOMES:
days without delirium | 5 days postoperative
  days
duration of delirium if it appear | 7 days postoperative
  days
severity of delirium | 7 days postoperative
  DRS-R-89
length of stay in the ICU | 3 days postoperative
  days
the length of stay in the hospital | 7 days postoperative
  days
the ICU mortality | 3 days postoperative
  number

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university hospitals, Cairo, Egypt